CLINICAL TRIAL: NCT03887624
Title: A Randomized, Parallel-group，Placebo-controlled, Double-blind Clinical Trial to Evaluate the Efficacy and Safety of Ethosuximide in Chinese Patients With Treatment-Resistant Depression.
Brief Title: Investigate the Clinical Responses of Ethosuximide in Patients With Treatment-Resistant Depression.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xu Yi, Doctor of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-716
Record Dates: First submitted 2019-03-02; First posted 2019-03-25 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder, Treatment-Resistant
Keywords: Depressive Disorder, Treatment-Resistant; ethosuximide
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Ethosuximide; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a double-blind and double-simulation design. In the course of clinical study, all subjects, researchers and evaluators are blind to grouping information. The results of the study are audited by blind state data. The placebos are administered in capsules with no difference in appearance, color, weight or odor from the positive drugs. Both subjects and drugs are coded blindly.
  In the study, the coding system for research drugs have an emergency blindness detection procedure, so as to quickly identify the drugs in emergency medical condition, without destroying the blind design of clinical research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Ethosuximide(2 weeks) + Escitalopram (4 weeks)
  Interventions: Drug: Ethosuximide; Drug: Escitalopram
- Control group (Placebo Comparator): Placebo(2 weeks)+Escitalopram(4 weeks)
  Interventions: Drug: Placebo; Drug: Escitalopram

INTERVENTIONS:
Drug: Ethosuximide — 2 times/day, take it orally after breakfast/dinner; take 500mg in the morning and 500mg in the evening on day1, 500mg in the morning and 750mg in the evening on day2, 750mg in the morning and 750mg in the evening on day3, 750mg in the morning and 1000mg in the evening on day4, 1000mg in the morning and 1000mg in the evening on day5, maintain this dose until the end of treatment for 2 weeks.
  Other Names: Zarontin
  Arms: Experimental group
Drug: Placebo — 2 times/day, take it orally after breakfast/dinner; take 500mg in the morning and 500mg in the evening on day1, 500mg in the morning and 750mg in the evening on day2, 750mg in the morning and 750mg in the evening on day3, 750mg in the morning and 1000mg in the evening on day4, 1000mg in the morning and 1000mg in the evening on day5, maintain this dose until the end of treatment for 2 weeks.
  Other Names: Placebo(for Ethosuximide)
  Arms: Control group
Drug: Escitalopram — 1 time/day, 20mg/day, take it orally after breakfast, take it for 4 weeks without interruption.
  Other Names: Lexapro

SUMMARY:
This study evaluates the efficacy and safety of ethosuximide in the treatment of refractory depressive disorder in adults. Half of participants will receive ethosuximide and escitalopram in combination, while the other half will receive a placebo and escitalopram.

DETAILED DESCRIPTION:
Ethosuximide is a inhibitor of low-voltage-sensitive T-type calcium channels(T-VSCCs). It has higher selectivity to T-VSCCs and can enter cerebrospinal fluid through the blood-brain barrier, inhibit T-VSCCs on the lateral habenular nucleus neurons, and then inhibit the cluster discharge of neurons, resulting in a rapid antidepressant effect.

ELIGIBILITY:
Inclusion criteria

1. Inpatient of both sexes are aged from 18 to 65 years;
2. Diagnosis of major depressive disorder(single or recurrent episodes) is made according to DSM-V(the fifth Edition of Diagnostic and Statistical Manual of Mental Disorders) criteria;
3. Subjects with previous or current depressive episodes did not response to two different antidepressants with recommended doses and adequate duration (maximum treatment dose of at least 6 weeks);
4. The subjects who will score more than or equal to 22 points on the MADRS scale at screening and baseline period;
5. The subjects who will score more than or equal to 3 points on the first clause of MADRS scale at screening and baseline period;
6. Subjects who will sign written informed consent and volunteer to participate in the clinical study.

Exclusion criteria

1. Diagnoses of other mental disorders (such as organic mental disorders, schizophrenia, bipolar and related disorders, anxiety disorders, obsessive-compulsive disorders and so on) are made according to DSM-V criteria;
2. Depressive episodes, such as depression caused by hypothyroidism, secondary to a systemic disease or an organic mental disorder caused by a neurological disease;
3. Subjects with a history of attempted suicide, or currently at high suicide risk, or with suicide behavior/attempt, or scoring more than or equal to 3 points on the 10th clause of MADRS scale;
4. Subject whose score of MADRS scale in baseline period will be 25% lower than that in screening period;
5. Subjects with a history of severe or poorly controlled cardiovascular, liver, kidney, blood, endocrine, respiratory diseases, etc;
6. Subjects with a history of epileptic seizures, except for a single febrile convulsion in children;
7. Researchers believe that the results of subjects' physical and laboratory examinations are clinically significant abnormalities in screening or baseline period. The following indicators exceed the following criteria: 1)ALT or AST levels are 1.5 times higher than the upper limit of laboratory normal values. 2)Thyroid Function are 1.1 times higher than the upper or lower limit of normal values. 3) Serum creatinine values are 1.1 times higher than the upper limit of normal values. 4)The levels of blood urea nitrogen are higher than the upper limit of normal values;
8. The result of electrocardiogram (ECG) is abnormal in screening or baseline period, such as male subjects with QTc interval (> 450 ms) and female subjects with QTc interval (> 470 ms) , and the researchers thought it is not suitable for selection;
9. Subjects could not swallow oral medicines or have a history of gastrointestinal surgery or any other diseases that may interfere with drug absorption, distribution, metabolism or excretion;
10. Monoamine oxidase inhibitors (MAOIs) are taken by subjects now or within 2 weeks before screening. Subjects who took antipsychotics, antidepressants or mood stabilizers before randomization and these drugs' cleaning phase had less than five half-lives. Subjects who took fluoxetine within 1 month before screening. Subjects who continue to take Chinese medicines with antidepressant effects specified in the instructions after signing informed consent.
11. Subjects who received modified electroconvulsive therapy (MECT) , transcranial magnetic stimulation (TMS), vagal nerve stimulation (VNS), or systematic psychotherapy within 3 months before screening;
12. Subjects with a history of allergies to two or more foods or drugs;
13. Subjects who addicted to alcohol or substances within 6 months before screening;
14. Prenatal, lactating, or reproductive women who had positive results of HCG tests before participating in the study; Male and female subjects will not take effective contraceptive measures or plan to be pregnant within 3 months after the study;
15. Subjects who participated in clinical research within 30 days before signing the informed consent form for this study;
16. According to the judgement of the researchers, other situations are not suitable for clinical research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale(MADRS） score | baseline and 43 days
  The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Usual cutoff points are: 0 to 6 - normal/symptom absent, 7 to 19 - mild depression, 20 to 34 - moderate depression, >34 - severe depression.
  Changes of MADRS score at therapeutic visit point compare with baseline.

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology-Self Report(QIDS-SR） score | baseline and 43 days
  The QIDS-SR is a psychological questionnaire used by clinicians to measure 16 factors across 9 different criterion domains for major depression. It is scored by summing the highest response in each of a set of questions relating to sleep, weight and psychomotor symptoms and then adding the remaining items. Scores range from 0 to 27 which may then be categorised as indicating none [0-5], mild [6-10], moderate [11-15], severe [16-20] and very severe [21-27] depressive symptoms.
  Changes of QIDS-SR score at therapeutic visit point compare with baseline.
Hamilton Anxiety Rating Scale(HAMA） score | baseline and 43 days
  The HAMA is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. Scores range from 0 to 56. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. Lastly, a score of 25 to 30 indicates a moderate to severe anxiety severity.
  Changes of HAMA score at therapeutic visit point compare with baseline.
MADRS score | baseline and 43 days
  Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6.
  Changes of individual score of MADRS at therapeutic visit point compare with baseline.
Young manic rating scale(YMRS） score | baseline and 43 days
  The Young Mania Rating Scale (YMRS) is an eleven-item multiple choice diagnostic questionnaire which psychiatrists use to measure the severity of manic episodes in children and young adults. The scores from each question are added together to form a total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms. Extremely high scores increase the risk of the child having bipolar disorder by a factor of 9, while extremely low scores decrease the risk by a factor of 10. A score of 13 or higher indicates a potential case of mania or hypomania, while a score of 21 or above indicates a probable case. The average score for children with mania is 25, while the average score for children with hypomania is 20.
  Changes of YMRS score at therapeutic visit point compare with baseline.
Efficiency after 2 and 4 weeks of treatment. | baseline, week 2 and week 4
  Efficiency means that the score of MADRS decreases by more than or equal to 50% compared with its baseline score.
Remission rate after 2 and 4 weeks of treatment. | baseline, week 2 and week 4
  Remission means that the total score of MADRS is less than 10.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Xu, Doctor of Medicine, Principal Investigator — Department of psychiatry, First Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Department of Psychiatry, the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sackeim HA. The definition and meaning of treatment-resistant depression. J Clin Psychiatry. 2001;62 Suppl 16:10-7. PMID 11480879
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Yang Y, Cui Y, Sang K, Dong Y, Ni Z, Ma S, Hu H. Ketamine blocks bursting in the lateral habenula to rapidly relieve depression. Nature. 2018 Feb 14;554(7692):317-322. doi: 10.1038/nature25509. PMID 29446381
- [Background] Cui Y, Yang Y, Ni Z, Dong Y, Cai G, Foncelle A, Ma S, Sang K, Tang S, Li Y, Shen Y, Berry H, Wu S, Hu H. Astroglial Kir4.1 in the lateral habenula drives neuronal bursts in depression. Nature. 2018 Feb 14;554(7692):323-327. doi: 10.1038/nature25752. PMID 29446379
- [Background] Sarkisova KY, Kuznetsova GD, Kulikov MA, van Luijtelaar G. Spike-wave discharges are necessary for the expression of behavioral depression-like symptoms. Epilepsia. 2010 Jan;51(1):146-60. doi: 10.1111/j.1528-1167.2009.02260.x. Epub 2009 Aug 8. PMID 19674046
- [Background] Cui Y, Hu S, Hu H. Lateral Habenular Burst Firing as a Target of the Rapid Antidepressant Effects of Ketamine. Trends Neurosci. 2019 Mar;42(3):179-191. doi: 10.1016/j.tins.2018.12.002. PMID 30823984

DOCUMENTS (3):
  • Study Protocol (2019-04-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03887624/Prot_004.pdf
  • Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03887624/SAP_003.pdf
  • Informed Consent Form (2019-04-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03887624/ICF_005.pdf